CLINICAL TRIAL: NCT02588573
Title: Overall Performance of a 1-day Silicone Hydrogel Lens When Habitual Soft Lens Wearers Are Refit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-61
Record Dates: First submitted 2015-10-22; First posted 2015-10-28 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etafilcon A (control) (Active Comparator): Subjects in each of the habitual wearing groups will be randomized to wear either the test or control lens in either the left or right eye.
  Interventions: Device: etafilcon A (control); Device: somofilcon A (test)
- Somofilcon A (test) (Active Comparator): Subjects in each of the habitual wearing groups will be randomized to wear either the test or control lens in either the left or right eye.
  Interventions: Device: etafilcon A (control); Device: somofilcon A (test)

INTERVENTIONS:
Device: etafilcon A (control) — contact lens
Device: somofilcon A (test) — contact lens

SUMMARY:
The objective of the study is to compare the overall subjective comfort profile over 8 hours of lens wear in two groups of habitual soft contact lens wearers (daily disposable hydrogel lenses and frequent replacement lenses) when refitted in to somofilcon A lenses.

DETAILED DESCRIPTION:
This will be a prospective, single day, randomized, double-masked, non-dispensing, contralateral study. Participants were recruited into one of two groups - participants who habitually wore etafilcon A: daily disposable hydrogel lenses and participants who habitually wore frequent replacement lenses (FREQ).

ELIGIBILITY:
Inclusion Criteria:

* A person is eligible for inclusion in the study if he/she:

  1. Is at least 17 years of age and has full legal capacity to volunteer;
  2. Has read and signed an information consent letter;
  3. Is willing and able to follow instructions and maintain the appointment schedule;
  4. Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual correction or the assigned study lenses;
  5. Habitually wears either etafilcon A lens or any frequent replacement contact lenses (as defined in 4.1.1);
  6. Habitually wear contact lenses with a power between -1.00 and -6.00D (Diopters) (inclusive) in both eyes;
  7. Demonstrates an acceptable fit with the study lenses;
  8. Is usually able to wear contact lenses for at least 8 hours per day.

Exclusion Criteria:

* A person will be excluded from the study if he/she:

  1. Is participating in any concurrent clinical or research study;
  2. Has any known active* ocular disease and/or infection;
  3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
  4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
  5. Has known sensitivity to the diagnostic substances (pharmaceuticals), such as fluorescein dye, or products to be used in the study;
  6. Is aphakic;
  7. Has undergone refractive error surgery.
  8. Has participated in the previous somfofilcon A study (ORE# 20893)

     * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Contact Lens Research
Locations (2):
- Canada (2):
  - Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario
  - University of Waterloo, Waterloo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 103 enrolled, 13 participants were not eligible due to screen failure. This reporting group includes 90 participants (180 eyes) belonging to 2 groups of 45 habitual wearers of either etafilcon A lens or frequent replacement lenses (FREQ). All participants were randomized to wear etafilcon A in one eye and somofilcon A in the fellow eye.
Units Other Than Participants: eyes
Groups:
- Habitual Etafilcon A Wearers: Habitual wearers of etafilcon A were randomized to wear etafilcon A lens in one eye and somofilcon A lens in the other eye for 8 hours during the contralateral study
- Habitual FREQ Wearers: Habitual wearers of other frequent replacement lenses (FREQ) were randomized to wear etafilcon A lens in one eye and somofilcon A lens in the other eye for 8 hours during the contralateral study.
Period: Overall Study
Arm/Group | Habitual Etafilcon A Wearers | Habitual FREQ Wearers
Started | 45; 90 eyes | 45; 90 eyes
Randomized Eye Etafilcon A | 45; 45 eyes | 45; 45 eyes
Randomized Eye Somofilcon A | 45; 45 eyes | 45; 45 eyes
Completed | 45; 90 eyes | 45; 90 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- Habitual Etafilcon A Wearers Wearing Etafilcon A/Somofilcon A: Habitual wearers of etafilcon A were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design for 8 hours during the study.
- Habitual FREQ Wearers Wearing Etafilcon A/Somofilcon A: Habitual wearers of frequent replacement lenses (FREQ) were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design for 8 hours during the study.
- Total: Total of all reporting groups
Arm/Group | Habitual Etafilcon A Wearers Wearing Etafilcon A/Somofilcon A | Habitual FREQ Wearers Wearing Etafilcon A/Somofilcon A | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Full Range); unit: years] | 25 [17 to 55] | 25 [17 to 63] | 25 [17 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective ratings for lens comfort of etafilcon A and somofilcon A. Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Habitual Etafilcon A Wearers Randomized to Etafilcon A: Habitual wearers of etafilcon A were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
  etafilcon A (control): contact lens
- Habitual Etafilcon A Wearers Randomized to Somofilcon A: Habitual wearers of etafilcon A were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
  somofilcon A (test): contact lens
- Habitual FREQ Wearers Randomized to Etafilcon A: Habitual wearers of frequent replacement lenses (FREQ) were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
  etafilcon A (control): contact lens
- Habitual FREQ Wearers Randomized to Somofilcon A: Habitual wearers frequent replacement lenses (FREQ) were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
  somofilcon A (test): contact lens
Arm/Group | Habitual Etafilcon A Wearers Randomized to Etafilcon A | Habitual Etafilcon A Wearers Randomized to Somofilcon A | Habitual FREQ Wearers Randomized to Etafilcon A | Habitual FREQ Wearers Randomized to Somofilcon A
Number analyzed (Participants) | 45 | 45 | 45 | 45
Number analyzed (eyes) | 45 | 45 | 45 | 45
units on a scale | 83 (17) | 77 (22) | 83 (14) | 83 (16)

2. Primary Outcome: Comfort Preference
Description: Lens preference in regards to comfort of etafilcon A and somofilcon A. Categories: Strongly prefer etafilcon A lens, slightly prefer etafilcon A lens, no preference, slightly prefer somofilcon A lens, strongly prefer somofilcon A lens
Time Frame: Baseline and 8 hours
Measure: Number; unit: participants
Groups:
- Habitual Etafilcon A Wearers - Baseline; Habitual Etafilcon A Wearers - 8hrs: Habitual wearers of etafilcon A were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
- Habitual FREQ Wearers - Baseline; Habitual FREQ Wearers - 8hrs: Habitual wearers of frequent replacement lenses (FREQ) were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
Arm/Group | Habitual Etafilcon A Wearers - Baseline | Habitual FREQ Wearers - Baseline | Habitual Etafilcon A Wearers - 8hrs | Habitual FREQ Wearers - 8hrs
Number analyzed (Participants) | 45 | 45 | 45 | 45
participants
  Strongly Prefer Etafilcon A Lens | 7 | 3 | 13 | 2
  Slightly Prefer Etafilcon A Lens | 14 | 10 | 11 | 16
  No Preference | 12 | 19 | 5 | 10
  Slightly Prefer Somofilcon A Lens | 10 | 11 | 9 | 8
  Strongly Prefer Somofilcon A Lens | 2 | 2 | 7 | 9

3. Primary Outcome: Bulbar Hyperemia
Description: Bulbar hyperemia examination using Efron scale 0-4, 0.5 steps, 0=normal, 4=severe.
Time Frame: Baseline and 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Habitual Etafilcon A Wearers Randomized to Etafilcon A; Habitual Etafilcon A Wearers Randomized to Somofilcon A: Habitual wearers of etafilcon A were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
- Habitual FREQ Wearers Randomized to Etafilcon A; Habitual FREQ Wearers Randomized to Somofilcon A: Habitual wearers of frequent replacement lenses (FREQ) were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
Arm/Group | Habitual Etafilcon A Wearers Randomized to Etafilcon A | Habitual Etafilcon A Wearers Randomized to Somofilcon A | Habitual FREQ Wearers Randomized to Etafilcon A | Habitual FREQ Wearers Randomized to Somofilcon A
Number analyzed (Participants) | 45 | 45 | 45 | 45
Number analyzed (eyes) | 45 | 45 | 45 | 45
units on a scale
  Baseline | 1.3 (0.4) | 1.3 (0.4) | 1.2 (0.4) | 1.2 (0.4)
  8 hours | 1.3 (0.4) | 1.3 (0.4) | 1.2 (0.4) | 1.2 (0.4)

4. Primary Outcome: Limbal Hyperemia
Description: Limbal hyperemia examination using Efron scale 0-4, 0.5 steps, 0=normal, 4=severe.
Time Frame: Baseline and 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Habitual Etafilcon A Wearers Randomized to Etafilcon A | Habitual Etafilcon A Wearers Randomized to Somofilcon A | Habitual FREQ Wearers Randomized to Etafilcon A | Habitual FREQ Wearers Randomized to Somofilcon A
Number analyzed (Participants) | 45 | 45 | 45 | 45
Number analyzed (eyes) | 45 | 45 | 45 | 45
units on a scale
  Baseline | 1.2 (0.5) | 1.2 (0.5) | 1.0 (0.4) | 1.0 (0.4)
  8 hours | 1.2 (0.4) | 1.3 (0.4) | 1.4 (0.5) | 1.3 (0.4)

5. Primary Outcome: Conjunctival Staining
Description: Conjunctival staining was graded in each quadrant with scale 0-4, 0.5 steps, 0=normal, 4=severe of four areas:
  N - Nasal, T - Temporal, S - Superior, I - Interior, C - Central
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Habitual Etafilcon A Wearers Randomized to Etafilcon A | Habitual Etafilcon A Wearers Randomized to Somofilcon A | Habitual FREQ Wearers Randomized to Etafilcon A | Habitual FREQ Wearers Randomized to Somofilcon A
Number analyzed (Participants) | 45 | 45 | 45 | 45
Number analyzed (eyes) | 45 | 45 | 45 | 45
units on a scale
  Nasal | 1.0 (0.8) | 1.1 (1.0) | 1.1 (1.0) | 1.4 (1.0)
  Temporal | 0.4 (0.5) | 1.1 (0.9) | 0.6 (0.6) | 1.4 (1.0)
  Superior | 0.3 (0.5) | 0.6 (0.8) | 0.2 (0.5) | 0.9 (0.8)
  Inferior | 0.6 (0.7) | 1.1 (1.0) | 0.6 (0.8) | 1.2 (1.2)

6. Primary Outcome: Visual Acuity
Description: High contrast visual acuity at high illumination was measured with each lens at each visit using a logMAR chart.
Time Frame: Baseline and 8 hours
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Habitual Etafilcon A Wearers Randomized to Etafilcon A | Habitual Etafilcon A Wearers Randomized to Somofilcon A | Habitual FREQ Wearers Randomized to Etafilcon A | Habitual FREQ Wearers Randomized to Somofilcon A
Number analyzed (Participants) | 45 | 45 | 45 | 45
Number analyzed (eyes) | 45 | 45 | 45 | 45
LogMAR
  Baseline | -0.05 (0.07) | -0.05 (0.09) | -0.07 (0.06) | -0.06 (0.08)
  8 hours | -0.06 (0.08) | -0.06 (0.10) | -0.07 (0.08) | -0.06 (0.08)

ADVERSE EVENTS:
Time Frame: 8 hours
Description: Adverse events will be monitored for during the follow-up visit.
Groups:
- Etafilcon A Lens (Control) Worn by Habitual Etafilcon A Grp; Somofilcon A Lens (Test) Worn by Habitual Etafilcon A Grp: Habitual wearers of etafilcon A were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
- Etafilcon A Lens (Control) Worn by Habitual FREQ Grp; Somofilcon A Lens (Test) Worn by Habitual FREQ Grp: Habitual wearers of frequent replacement lenses (FREQ) were randomized to wear somofilcon A lens (test) and etafilcon A lens (control) in a contralateral design.
Arm/Group | Etafilcon A Lens (Control) Worn by Habitual Etafilcon A Grp | Somofilcon A Lens (Test) Worn by Habitual Etafilcon A Grp | Etafilcon A Lens (Control) Worn by Habitual FREQ Grp | Somofilcon A Lens (Test) Worn by Habitual FREQ Grp
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other